CLINICAL TRIAL: NCT07354308
Title: A Study to Evaluate the Efficacy of an Avocado Dietary Supplement to Support Healthy Weight and Blood Glucose Management
Brief Title: Study to Evaluate the Efficacy of an Avocado Dietary Supplement
Acronym: METAVO-ONE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SP Nutraceuticals Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20710
Record Dates: First submitted 2025-12-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Metabolic Health; Insulin Resistance
Keywords: Weight Management; Glucose Metabolism; avocado
MeSH Terms: conditions — Overweight; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metavo Supplement Group (Experimental): Participants in this group will receive the Metavo dietary supplement for 16 weeks.
  Interventions: Dietary Supplement: Metavo Supplement
- Placebo Group (Placebo Comparator): Participants in this group will receive placebo capsules that are visually matched to the Metavo supplement for 16 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Metavo Supplement — Participants will take 8 Intervention capsules per day (4 in the morning, 4 in the afternoon)
  Arms: Metavo Supplement Group
Dietary Supplement: Placebo — Participants will take 8 placebo capsules per day (4 in the morning, 4 in the afternoon)
  Arms: Placebo Group

SUMMARY:
This 16-week, randomized, triple-blinded, placebo-controlled study evaluates the effects of an avocado dietary supplement (Metavo) on healthy weight and blood glucose management in overweight adults. The study includes body measurements, questionnaires, blood tests, and CGM monitoring to assess metabolic outcomes and participant-reported perceptions of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be aged between 18 and 70 years of age
* Be classified as overweight or obese with a BMI of ≥25.0 and ≤32 kg/m2.
* Have a stable weight defined as <10% change in body weight in three months prior to the study start date.
* Willing to follow the provided diet and exercise guidelines.
* Willing to not consume avocados throughout the trial and for two weeks prior to Baseline
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Willing to stop any products, any prescription medication, or supplements that target weight management, blood sugar control, and/or aim to improve insulin during the test period.
* Willing to avoid introducing any new products or any new forms of prescription medication or supplements that target weight management, blood sugar control, and/or aim to improve insulin during the test period.
* Not currently partaking in another research study and will not be partaking in any other research study for the next 16 weeks and at any point during this study's duration.
* Must have someone available to take front and side profiles of the torso.
* Must have a smart phone or camera capable of taking photos of the torso.
* Resides in the United States.

Exclusion Criteria:

* Anyone with diagnosed Type I or Type II diabetes.
* Allergic to avocados
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive
* Anyone unwilling to follow the study protocol.
* Has stopped using hormonal birth control in the past month.
* Anyone with a history of substance abuse.
* Anyone who is currently a smoker or has been a smoker in the past 6 months.
* Anyone with chronic health conditions that could impact participation in the study, such as oncological, psychiatric, metabolic, hypertension, or cardiovascular disorders, cancer, autoimmune disease, HIV, Hepatitis B, and/or C, kidney and/or liver, gastrointestinal, gastroesophageal reflux, blood/bleeding disorders, gout, or mental health disorders.
* Anyone who has had any major illness in the last 3 months.
* Anyone who drinks heavily (i.e., 8 or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men).
* Current use of prescribed medications as listed below: Weight loss prescription medication (within 3 months of baseline). Anticoagulants and coagulants (within 4 weeks of baseline).
* Anyone who has used any cannabis products (medical or recreational) in the past month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass | Baseline through Week 16
  Measured via Withings Smart Scale. Participants will weigh themselves daily for 3 consecutive days each week. If the first two values are similar, their average is used. If they differ by ≥10 lbs, the third value is used to determine the average.
Change in Average Blood Glucose | 2 weeks before Baseline and Weeks 14-16
  Change in average blood glucose levels measured using a Continuous Glucose Monitor (CGM). Average glucose will be calculated over each time period and the change from pre-baseline to Weeks 14-16 will be reported.
Change in Hemoglobin A1C (HbA1C) | Baseline and Week 16
  Assessed via blood samples at Labcorp or via home phlebotomy.
Change in Fasting Insulin | Baseline and Week 16
  Assessed via blood samples at Labcorp or via home phlebotomy.
Change in Lipid Panel | Baseline and Week 16
  Includes Cholesterol, LDL, VLDL, HDL, and triglycerides. Measured via Labcorp or home phlebotomy.
Change in hs-CRP | Baseline and Week 16
  High-sensitivity C-reactive protein measured via Labcorp or home phlebotomy.
Change in Fasting GLP-1 Levels | Baseline and Week 16
  Only measured in the home phlebotomy subgroup using InterScience Institute lab testing.
Change in Waist Circumference | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Measured with a tape measure.
Change in Time in Range (TIR) | 2 weeks before Baseline and Weeks 14-16
  Change in percentage of time that glucose levels are within the target range, measured using a CGM. TIR will be computed as the percentage of total CGM readings within the target range during the specified time periods.
Change in Time Below Range (TBR) | 2 weeks before Baseline and Weeks 14-16
  Change in percentage of time that glucose levels are below the target range, measured using a CGM. TBR will be calculated as the percentage of total CGM readings below the target range.
Change in Time Above Range (TAR) | 2 weeks before Baseline and Weeks 14-16
  Change in percentage of time that glucose levels are above the target range, measured using a CGM. TAR will be calculated as the percentage of total CGM readings above the target range.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Evaluated using the Short Form-12 (SF-12) questionnaire.
Change in Physical Activity | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Evaluated using the Godin Leisure-Time Exercise Questionnaire (GLTE).
Change in Eating Habits | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Evaluated using the Three-Factor Eating Questionnaire - Revised 21 (TFEQ-R21).
Change in Food Cravings | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Evaluated using the Food Craving Questionnaire - Trait reduced (FCQ-T reduced).
Change in Self-Reported Mood, Energy, and Health | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Participants report changes in energy levels, weight perception, mood, and general well-being.
Change in Total Muscle Mass (kg) | Weekly from Baseline to Week 16
  Total skeletal muscle mass measured in kilograms using a Withings smart scale via Bioelectrical Impedance Analysis (BIA).
Change in Total Body Fat Mass (kg) | Weekly from Baseline to Week 16
  Total weight of body fat measured in kilograms using a Withings smart scale via Bioelectrical Impedance Analysis (BIA).
Change in Bone Mass (kg) | Weekly from Baseline to Week 16
  Estimated weight of bone mineral content in kilograms, measured using a Withings smart scale via Bioelectrical Impedance Analysis (BIA).
Change in Total Lean Mass (kg) | Weekly from Baseline to Week 16
  Total fat-free mass (including muscle, bone, and water) measured in kilograms using a Withings smart scale via Bioelectrical Impedance Analysis (BIA).
Change in Total Body Water Percentage (%) | Weekly from Baseline to Week 16
  Total body water as a percentage of total body weight, measured using a Withings smart scale via Bioelectrical Impedance Analysis (BIA).
Change in Visceral Fat Index | Weekly from Baseline to Week 16
  An indexed score representing the amount of visceral fat (the fat surrounding internal organs) measured via a Withings smart scale. This index typically ranges from 1 to 20, where higher scores indicate higher visceral fat levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States